CLINICAL TRIAL: NCT02010164
Title: THE EFFECT OF COQ10 SUPPLEMENTATION ON FOLLICULAR CELLS' BIOLOGY/PROPERTIES IN ELDERLY IVF PATIENTS
Brief Title: CoQ10 Treatment to Improve Fertility in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoQ10follicle
Record Dates: First submitted 2013-11-26; First posted 2013-12-12 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Reproductive Physiological Phenomena
Keywords: Reproductive aging; Mitochondria
MeSH Terms: interventions — coenzyme Q10

ARMS (3):
- Old-CoQ10 (Experimental)
  Interventions: Dietary Supplement: Co-enzyme Q10
- Old (No Intervention)
- Young (No Intervention): Young less than 33 years old participants

INTERVENTIONS:
Dietary Supplement: Co-enzyme Q10 — 600mg for 3 months
  Arms: Old-CoQ10

SUMMARY:
Delaying first childbirth is a progressive trend in the developed societies. Several theories tried to explain the reproductive aging, in purpose to hasten it. One of the theories include mitochondrial dysfunction with aging. In this study we will investigate the potential of treating elderly IVF patients with CoQ10, a mitochondrial stimulator, to improve follicle cells' properties.

DETAILED DESCRIPTION:
Over the past 4 decades, because of cultural and social changes, women in the developed world have significantly delayed childbirth. It is well known that fertility decreases with age and that live birth rates in women over the age of 35 are significantly lower both naturally and with assisted reproduction compared to those in women under the age of 35. The decline in live birth rate reflects an increase in oocyte aneuploidy that leads to reduced embryo quality as well as an increased incidence of miscarriages and birth defects, most prominently Down's syndrome (trisomy 21). There is evidence that older infertility patients have abnormal oocyte mitochondrial activity and reduced production of ATP. The meiotic spindle, crucial for normal chromosome segregation, may not be formed properly in the absence of appropriate ATP levels. Altered spindles may result in aneuploid embryos, which implant poorly or not at all.

Coenzyme Q10 (CoQ10) is a vitamin-like antioxidant, essential for proper function of mitochondrial respiratory chain. It has been shown that there is a decrease level of CoQ10 in several tissues with aging (like muscle). We suggest that one possible explanation for altered oocyte mitochondrial function may be diminished CoQ10 substrate availability or utilization as a function of aging. The oocytes, and in fact the pre-granulosa cells which give rise to the granulosa (GC) and cumulus cells (CC), are unique in the body since there is no cell division for many years. Therefore, in older women, the oocytes and GCs in primordial follicles will have been exposed to low levels of radical oxygen species produced by mitochondrial respiration over decades, resulting in possible cumulative damage to mitochondria and DNA. Decreased availability of CoQ10 would contribute to reduced antioxidant activity and decreased ATP production by the mitochondria in the oocyte. In addition, compromised mitochondrial function in GCs can effect steroid hormone production, as steroidogenesis is initiated in the inner mitochondrial membrane. Thus, a vicious circle is created by which decreased CoQ10 bioavailability with advanced age could adversely affect meiosis and further developmental competence of gametes.

In our mice model, we demonstrated mitochondrial dysfunction in oocytes from aged dams. Of importance, we found that many of these mitochondrial abnormalities could be partially or completely corrected by maternal supplementation with CoQ10, translated into significant increase in litter size of old -treated females. We could demonstrate also "normalization" of viability and function of CC (that "nourish" oocyte) by CoQ10 supplementation. The aim of the proposed project is to investigate CoQ10 levels and CC function in women with aging and the potential of CoQ10 treatment to improve follicular function, and as a result, improve oocyte quality. If intra-follicular CoQ10 levels are shown to decrease with maternal aging, nutritional supplementation with CoQ10 can become the future "folic acid" for improving reproductive outcomes in older women and not just those with infertility issues.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old patients undergoing IVF/ICSI

Exclusion Criteria:

* BMI>35
* already treated with CoQ10
* HCV carriers
* had experimental treatment in the last 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Follicular fluid CoQ10 levels | Change in CoQ10 levels before and after 90 days of treatment
cumulus cells function | Change in cumulus cells function before and after 90 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Israel